CLINICAL TRIAL: NCT02309138
Title: Comparison of Two Screening Strategies for Gestational Diabetes (GDM2)
Acronym: GDM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esa M Davis, MD MPH FAAFP (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Esa M Davis, MD MPH FAAFP, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: PRO14070556; R01HD079647 (NIH)
Record Dates: First submitted 2014-11-25; First posted 2014-12-05 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Gestational Diabetes; Pregnancy; Glucose Intolerance
Keywords: gestational diabetes screening; Carpenter Coustan Criteria; IADPSG criteria; Large for gestational age birth weight
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 3 hour 100 gm OGTT (CC Criteria) (Active Comparator): Gestational diabetes screening with fasting 3 hour 100 gm. Receive a fasting 3 hour 100 gram oral glucose tolerance test and are diagnosed based on the Carpenter Coustan Criteria: a 50 gm Glucose tolerance test of >130 + fasting 3 hour 100 gram oral glucose tolerance test with two or more values greater than the following diagnostic threshold: Fasting 95, 1-hour 180, 2-hour 155, or 3 hour 140 mg/dL . A positive criteria will be diagnostic for gestational diabetes.
  Interventions: Diagnostic Test: Gestational diabetes screening with fasting 3 hour 100 gm
- 2 hr 75 gm OGTT (IADPSG Criteria) (Active Comparator): Gestational diabetes screening with fasting 2 hour 75g. Receive a fasting 2 hour 75 gm oral glucose tolerance test and diagnosed based on the IADPSG which is if one or more values exceed the following diagnostic threshold: Fasting 92, 1-hour 180, or 2-hour 153 mg/dL.
  Interventions: Diagnostic Test: Gestational diabetes screening with fasting 2 hour 75g

INTERVENTIONS:
Diagnostic Test: Gestational diabetes screening with fasting 3 hour 100 gm — Participants receive fasting 3 hour 100 gm oral glucose tolerance test
  Arms: 3 hour 100 gm OGTT (CC Criteria)
Diagnostic Test: Gestational diabetes screening with fasting 2 hour 75g — Participants receive fasting 2 hour 75 gm oral glucose tolerance test
  Arms: 2 hr 75 gm OGTT (IADPSG Criteria)

SUMMARY:
This is a single site blinded RCT of 920 pregnant women with singleton gestation designed to compare the Carpenter-Coustan and IADPSG criteria for diagnosing gestational diabetes. Maternal metabolic profiles and infant growth will be assessed at randomization and at one year postpartum.

DETAILED DESCRIPTION:
Impaired glucose metabolism (gestational diabetes (GDM) and mild hyperglycemia) that occurs during pregnancy is associated with an increased risk for pregnancy complications and is also an early indication of long-term metabolic dysfunction leading to diabetes and cardiovascular disease. In the US, GDM is diagnosed using a two-step screening and diagnostic approach. The International Association of Diabetes and Pregnancy Study Group (IADPSG) proposed a one-step diagnostic approach that broadens the definition of GDM by lowering the cutoff values to include women with milder forms of hyperglycemia, who would have screened normal under the current two-step approach. The goal of these recommendations is better identification of women at risk for pregnancy complications and long-term metabolic dysfunction, but it results in a significant increase in the prevalence of GDM. The NIH GDM Consensus Development Conference committee does not recommend changing from the current two-step screening/diagnostic approach to the IADPSG one-step diagnostic approach without trials demonstrating that increasing the number of women diagnosed as having GDM results in better outcomes. We aim to 1) conduct a "real world" randomized controlled trial (RCT) to determine differences in short-term perinatal health outcomes between the two predominant GDM screening approaches, and 2) prospectively follow the mothers to examine their metabolic risk profiles and the growth of their infants at 1 year postpartum. Based on a pilot study, we propose a single site blinded RCT of 920 pregnant women ages 18-45 years without a diagnosis of diabetes, with a singleton pregnancy (18-24 wks gestation). Participants will have a non-fasting 1 hour 50 gm glucose challenge test (GCT) performed between 24-28 weeks' gestation. Women with 50 gm GCT results < 200 mg/dL will be randomized to receive either a fasting 2 hour 75 gm oral glucose tolerance test (OGTT) or a 3 hour 100 gm OGTT. GDM will be diagnosed using the IADPSG criteria for women receiving the 75 gm OGTT and Carpenter-Coustan criteria for women receiving the 100 gm. Participants and their physicians will be informed of the diagnosis of GDM, but blinded to the specific test results and diagnostic criteria. Participants with GDM will receive treatment from their primary provider. Questionnaires will be used to assess participants' and physicians' views on GDM testing. Metabolic profiles will be assessed at randomization and at a year postpartum. The primary outcome measure is large-for-gestational age fetal growth. The rationale for this RCT is that this is a unique opportunity to compare the two methods. At the end of the study, we will know whether women diagnosed at lower glucose levels with the IADPSG criteria are more likely to have adverse perinatal outcomes. We hypothesize that using IADPSG diagnostic criteria will result in greater detection of women with impaired glucose metabolism and treating these women will reduce adverse perinatal outcomes and prevent long-term metabolic dysfunction. This study will provide level A data for endorsing universal screening guidelines for GDM by major organizations and implementation into clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 18-24 weeks of gestation
* Singleton gestation
* Planning to deliver at Magee-Womens Hospital, Pittsburgh, Pennsylvania

Exclusion Criteria:

* Preexisting type 1 or 2 diabetes
* Diabetes diagnosed at less than 24 weeks gestational age (GA)
* Multiple gestations ( e.g. twins or triplets)
* Hypertension requiring medications
* Corticosteroid (IM, oral or IV) use in the 30 days prior to enrollment
* Major congenital anomaly with anticipated preterm delivery due to maternal or fetal indications < 28 wks GA
* Inability to complete the glucose testing before 30 completed weeks GA
* Advanced HIV( on medications that cause hyperglycemia), severe liver disease, gastric bypass surgery or other illness/surgeries that preclude them from drinking the glucola solution.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 921 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esa M Davis, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed and the investigators have published the main manuscripts regarding the outcomes of the trial. De-identified data will be made available by request, review and approval of the investigators and the institution regulatory committee.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared in the appropriate time frame required by policy.
Access Criteria: An application and review process will be implemented for accessing data.

REFERENCES:
- [Background] Abebe KZ, Scifres C, Simhan HN, Day N, Catalano P, Bodnar LM, Costacou T, Matthew D, Illes A, Orris S, Duell J, Ly K, Davis EM. Comparison of Two Screening Strategies for Gestational Diabetes (GDM2) Trial: Design and rationale. Contemp Clin Trials. 2017 Nov;62:43-49. doi: 10.1016/j.cct.2017.08.012. Epub 2017 Aug 18. PMID 28823926
- [Derived] Scifres CM, Davis EM, Orris S, Costacou T, Lalama C, Abebe KZ, Catalano P. Metabolic factors and perinatal outcomes among pregnant individuals with mild glucose intolerance. Diabetes Res Clin Pract. 2024 Oct;216:111830. doi: 10.1016/j.diabres.2024.111830. Epub 2024 Aug 17. PMID 39159865
- [Derived] Davis EM, Abebe KZ, Simhan HN, Catalano P, Costacou T, Comer D, Orris S, Ly K, Decker A, Mendez D, Day N, Scifres CM. Perinatal Outcomes of Two Screening Strategies for Gestational Diabetes Mellitus: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jul 1;138(1):6-15. doi: 10.1097/AOG.0000000000004431. PMID 34259458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women were recruited from June 2015 to February 2019 from 10 obstetrical clinics affiliated with Magee Women's Hospital in Pittsburgh,Pennsylvania
Groups:
- 2 hr 75 gm OGTT (IADPSG Criteria): Gestational diabetes screening with fasting 2 hour 75g. Receive a fasting 2 hour 75 gm oral glucose tolerance test and diagnosed based on the International Association of the Diabetes in Pregnancy Study Group (IADPSG) which is if one or more values exceed the following diagnostic threshold: Fasting 92, 1-hour 180, or 2-hour 153 mg/dL.
  Gestational diabetes screening with fasting 2 hour 75g: Participants receive fasting 2 hour 75 gm oral glucose tolerance test
Period: Overall Study
Arm/Group | 3 Hour 100 gm OGTT (CC Criteria) | 2 hr 75 gm OGTT (IADPSG Criteria)
Started | 460 | 461
Completed | 412 | 443
Not Completed | 48 | 18
Not completed — Withdrawal by Subject | 44 | 15
Not completed — Protocol Violation | 4 | 2
Not completed — delivered before visit 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Hour 100 gm OGTT (CC Criteria) | 2 hr 75 gm OGTT (IADPSG Criteria) | Total
Number analyzed (Participants) | 460 | 461 | 921
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (5.1) | 28.6 (5.3) | 28.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 460 | 461 | 921
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 443 | 445 | 888
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 18 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 161 | 139 | 300
  White | 249 | 261 | 510
  More than one race | 26 | 27 | 53
  Unknown or Not Reported | 14 | 14 | 28
pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m2] — Population: participant data missing
  kg/m2
    number analyzed (Participants) | 399 | 428 | 827
    (all) | 26.6 (6.8) | 26.9 (7.2) | 26.8 (7.0)
Glucose Challenge 50 gm test [Mean (Standard Deviation); unit: mg/dl] | 104.7 (27.7) | 107.8 (28.9) | 106.2 (28.3)
previous history of gestational diabetes [Count of Participants; unit: Participants] — Population: participant missing data
  Participants
    number analyzed (Participants) | 399 | 429 | 828
    (all) | 8 | 14 | 22
First degree family history of diabetes [Count of Participants; unit: Participants] — Population: participant missing data
  Participants
    number analyzed (Participants) | 393 | 415 | 808
    (all) | 97 | 103 | 200

OUTCOME MEASURES:

1. Primary Outcome: Large for Gestational Age (LGA) Infant
Description: birth weight equal to or greater than the 90th percentile for gestational age and sex
Time Frame: at time of delivery
Measure: Count of Participants; unit: Participants
Groups:
- Overall IADPSG Arm: Participants randomized into the IADPSG arm
- Overall Carpenter Coustan: Participants randomized in the the Carpenter Coustan arm
- IADPSG With no GDM: Participants diagnosed as having no GDM by the IADPSG criteria.
- Carpenter Coustan With no GDM: Participants diagnosed as having no GDM by the Carpenter Coustan criteria
Arm/Group | Overall IADPSG Arm | Overall Carpenter Coustan | IADPSG With no GDM | Carpenter Coustan With no GDM
Number analyzed (Participants) | 443 | 412 | 364 | 377
Participants | 34 | 35 | 28 | 34
Statistical Analysis 1: Comparison: Overall IADPSG Arm vs Overall Carpenter Coustan; Co-primary hypotheses #1: women diagnosed using the IADPSG criteria will have lower rates of large-for-gestational age infants compared to those diagnosed using the Carpenter-Coustan criteria; Test type: Superiority; p = 0.668, Regression, Logistic — Each co-primary hypothesis was tested at the 2.5% significance level; In the ITT, logistic regression was used to quantify the probability of large-for-gestational age as a function of the study arm and clinic type; Risk Ratio (RR) = 0.903, 97.5% CI 2-sided [0.538 to 1.516] — A relative risk < 1 represents a benefit in the direction of the IADPSG group, while a value > 1 represents a benefit towards the CC group
Statistical Analysis 2: Comparison: IADPSG With no GDM vs Carpenter Coustan With no GDM; Co-primary hypothesis #2: women classified as "no gestational diabetes" by the IADPSG criteria will have lower rates of large-for-gestational age infants compared to those classified in the Carpenter-Coustan criteria; Test type: Superiority; p = 0.853, Regression, Logistic — Each co-primary hypothesis was tested at the 2.5% significance level; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.853, 97.5% CI 2-sided [0.493 to 1.475]

2. Secondary Outcome: Cesarean Delivery
Description: the delivery of a baby through a surgical incision in the mother's abdomen and uterus
Time Frame: at delivery (approximately 40 weeks' gestation)
Measure: Count of Participants; unit: Participants
Groups:
- Overall Carpentar-Coustan Arm: Participants randomized in the the Carpenter Coustan arm
- IADPSG Criteria w/ No GDM: Participants randomized in the the IADPSG arm w "No GDM" classification
- CC Criteria w/ No GDM: Participants randomized in the the Carpenter Coustan arm w/ "No GDM" classification
Arm/Group | Overall IADPSG Arm | Overall Carpentar-Coustan Arm | IADPSG Criteria w/ No GDM | CC Criteria w/ No GDM
Number analyzed (Participants) | 449 | 423 | 365 | 377
Participants | 131 | 118 | 101 | 101
Statistical Analysis 1: Comparison: Overall IADPSG Arm vs Overall Carpentar-Coustan Arm; Test type: Superiority; p = 0.6669, Regression, Logistic; Risk Ratio (RR) = 1.046, 95% CI 2-sided [0.847 to 1.291]
Statistical Analysis 2: Comparison: IADPSG Criteria w/ No GDM vs CC Criteria w/ No GDM; Test type: Superiority; p = 0.8394, Regression, Logistic; Risk Ratio (RR) = 1.033, 95% CI 2-sided [0.816 to 1.307]

3. Secondary Outcome: Maternal Composite Morbidity
Description: maternal pre-eclampsia, 3rd or 4th degree vaginal lacerations, post-partum hemorrhage
Time Frame: at delivery (approximately 40 weeks' gestation)
Measure: Count of Participants; unit: Participants
Groups:
- Carpenter Coustan With no GDM: Participants diagnosed as having no GDM by the CC criteria
Arm/Group | Overall IADPSG Arm | Overall Carpenter Coustan | IADPSG With no GDM | Carpenter Coustan With no GDM
Number analyzed (Participants) | 442 | 425 | 365 | 379
Participants | 77 | 75 | 62 | 63
Statistical Analysis 1: Comparison: Overall IADPSG Arm vs Overall Carpenter Coustan; Test type: Superiority; p = 0.9335, Regression, Logistic; Risk Ratio (RR) = 0.987, 95% CI 2-sided [0.740 to 1.318]
Statistical Analysis 2: Comparison: IADPSG With no GDM vs Carpenter Coustan With no GDM; Test type: Superiority; p = 0.9260, Regression, Logistic; Risk Ratio (RR) = 1.022, 95% CI 2-sided [0.742 to 1.407]

4. Secondary Outcome: Neonatal Composite Morbidity
Description: 1) hypoglycemia: blood glucose < 40mg/dl); 2) hyperbilirubinemia requiring treatment, clinical jaundice; 3)hyperinsulinemia- measured with c peptide level from venous cord blood; 4) still birth- absence of fetal heart tones before delivery, 5) birth trauma= Shoulder dystocia/brachial plexus injuries.
Time Frame: 7 days after birth
Measure: Count of Participants; unit: Participants
Groups:
- IADPSG Without GDM: Participants diagnosed as having no GDM by IADPSG criteria
- Carpenter Coustan Without GDM: Participants diagnosed as having no GDM with the Carpenter Coustan criteria
Arm/Group | 2 hr 75 gm OGTT (IADPSG Criteria) | 3 Hour 100 gm OGTT (CC Criteria) | IADPSG Without GDM | Carpenter Coustan Without GDM
Number analyzed (Participants) | 442 | 425 | 365 | 379
Participants | 83 | 57 | 57 | 48
Statistical Analysis 1: Comparison: 2 hr 75 gm OGTT (IADPSG Criteria) vs 3 Hour 100 gm OGTT (CC Criteria); Test type: Superiority; p = 0.0322, Regression, Logistic; Risk Ratio (RR) = 1.400, 95% CI 2-sided [1.027 to 1.909]
Statistical Analysis 2: Comparison: IADPSG Without GDM vs Carpenter Coustan Without GDM; Test type: Superiority; p = 0.2643, Regression, Logistic; Risk Ratio (RR) = 1.233, 95% CI 2-sided [0.864 to 1.760]

ADVERSE EVENTS:
Time Frame: Adverse events timeframe in which data were collected was from the time of enrollment of the first participants to the final participant 12 month F/U (~ 5 years). However, adverse event data on each participants was collected within 48 hours of the requirement to fast prior to lab work done for the study and any serious adverse events were collected between study visit 1 and 2 and visit 2and delivery, and determined if related to the study procedures.
Arm/Group | 3 Hour 100 gm OGTT (CC Criteria) | 2 hr 75 gm OGTT (IADPSG Criteria)
All-Cause Mortality (participants affected / at risk) | 0/460 | 0/461
Serious Adverse Events (participants affected / at risk) | 17/460 | 2/461
Other Adverse Events (participants affected / at risk) | 154/460 | 56/461
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Hour 100 gm OGTT (CC Criteria) (N=460) | 2 hr 75 gm OGTT (IADPSG Criteria) (N=461)
Hypoglycemia (Metabolism and nutrition disorders) | 12 (12) | 1 (1) — < 40-30 mg/dl; <2.2-1.7 mol/L
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) — < 30 mg/dl; <1.7 mol/L, life threatening consequences; seizures
migraine headache (Nervous system disorders) | 1 (1) | 0 (0) — went to Emergency room and as tx and released.
heavy vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Admitted to hospital with vaginal bleeding due to placenta previa
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Pt had spontaneous premature rupture of members right during study visit
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 Hour 100 gm OGTT (CC Criteria) (N=460) | 2 hr 75 gm OGTT (IADPSG Criteria) (N=461)
nausea (Metabolism and nutrition disorders) | 58 (58) | 20 (20)
dizziness (Nervous system disorders) | 22 (23) | 4 (4)
vomiting (Gastrointestinal disorders) | 28 (30) | 12 (12)
Malaise (General disorders) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 4 (4)
Other (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 70 (72) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT02309138/SAP_000.pdf
  • Study Protocol (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02309138/Prot_001.pdf